CLINICAL TRIAL: NCT04025372
Title: INTREPId (INTermediate Risk Erection PreservatIon Trial): A Randomized Trial of Radiation Therapy and Darolutamide for Prostate Cancer
Brief Title: INTREPId (INTermediate Risk Erection PreservatIon Trial)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bayer (Industry); Decipher Biosciences (Unknown)
Responsible Party: Principal Investigator, Martin T. King, MD, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-202
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Gonadotropin-Releasing Hormone; Radiotherapy; darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bicalutamide+GnRH Agonist+Radiation Therapy (Experimental): * Bicalutamide is administered orally on a daily basis
  * GnRH Agonist as prescribed
  * Radiation therapy is administered starting 4-16 weeks after ADT
  Interventions: Drug: Bicalutamide; Drug: GnRH Agonist; Radiation: Radiation Therapy
- Darolutamide+Radiation Therapy (Experimental): * Darolutamide is administered orally twice daily
  * Radiation therapy is administered starting 4-16 weeks after Darolutamide
  Interventions: Radiation: Radiation Therapy; Drug: Darolutamide

INTERVENTIONS:
Drug: Bicalutamide — Bicalutamide is categorized as an antiandrogen. Antiandrogens are substances that block the effects of testosterone. Cancer of the prostate depends on the male hormone testosterone for its growth. If the amount of testosterone is reduced it is possible to slow down or shrink the cancer.
  Arms: Bicalutamide+GnRH Agonist+Radiation Therapy
Drug: GnRH Agonist — In men, GnRH agonists cause the testicles to stop making testosterone. Some GnRH agonists are used to treat prostate cancer.
  Arms: Bicalutamide+GnRH Agonist+Radiation Therapy
Radiation: Radiation Therapy — Radiation Therapy is a cancer treatment that uses high doses of radiation to kill cancer cells and shrink tumors.
Drug: Darolutamide — Darolutamide belongs to a class of drugs called androgen receptor inhibitors. In the body, these agents compete with androgens for binding to the androgen receptor, which reduces the ability of androgens to promote the growth of prostate cancer cells
  Arms: Darolutamide+Radiation Therapy

SUMMARY:
This research study is comparing the use of a new form of hormonal therapy used with radiation as a possible treatment for intermediate risk prostate cancer. More specifically, this research would help determine whether this new form of hormonal therapy is as effective as the standard hormone therapy while also preserving erectile function.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means that the drug is being studied.

In this research study, the investigators are looking at whether the novel form of hormonal therapy, called Darolutamide, when paired with radiation therapy will provide the same quality of care as the current standard treatments available for men with this type of cancer. Darolutamide prevents testosterone from signaling throughout the body. Although studies have shown that Darolutamide has activity in more advanced forms of prostate cancer, the activity of Darolutamide is unknown in intermediate risk prostate cancer treated with radiation therapy. The U.S. Food and Drug Administration (FDA) has not approved Darolutamide as a treatment for any disease.

The current standard of care treatments available to men with this type of cancer are radiation therapy with or without androgen deprivation therapy (ADT) involving a gonadotropin releasing hormone agonist plus bicalutamide (both FDA-approved) or surgery. ADT works by depriving the body of testosterone which "feeds" prostate cancer cells and weakens prostate cancer cells from repairing damage caused by radiation therapy.

In addition, the investigator will be assessing erectile function at baseline, during and after treatment to determine if short-term erectile function can be preserved without sacrificing long-term disease control.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma by biopsy within 1 year (365 days) from registration. The most recent biopsy will determine eligibility
* National Cancer Center Network (NCCN) intermediate risk prostate cancer, defined as clinical T2b-T2c, Gleason 7, or PSA 10-20 ng/mL. Patients who only have radiographic evidence of T3 disease (i.e. extracapsular extension, or seminal vesical invasion radiographically) will not be excluded.
* Able to characterize the number of unfavorable intermediate risk factors below:

  * 2-3 intermediate risk factors

    * T2b-T2c
    * Gleason 7
    * PSA 10-20 ng/mL
  * Gleason 4+3 disease
  * Percent positive cores ≥ 50%
* Tissue available for submission for Decipher genomic score from archived tissue. Patients who had tissue sent to Decipher but did not have sufficient tissue for processing will not be excluded. Patients who already have a Decipher score must present official report documentation.
* Able to undergo radiation therapy with curative intent
* Age ≥ 18 at the time of consent.
* Demonstrate adequate organ function (hematologic, renal, hepatic) within 3 months of registration
* System Laboratory Value
* Hematological:

  * Platelet count (plt) ≥ 100,000/ µL
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Absolute neutrophil count (ANC) ≥ 1000 cells/µL
* Renal:

  * Glomerular filtration rate (GFR) ≥ 45 mL/min

    * CKD-EPI equation will be used to calculate GFR
* Hepatic and Other:

  * Bilirubin ≤ 1.5 × upper limit of normal (ULN)

    * In subjects with Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin; if direct bilirubin is ≤1.5 × ULN, subject may be eligible
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
  * Serum Albumin > 3.0 g/dL
  * Serum potassium ≥ 3.5 mmol/L
* Endocrine:

  * Testosterone ≥ 150 ng/dL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Good erectile function, as assessed by 'firm enough for masturbation or foreplay' or 'firm enough for intercourse' response to the question "How would you describe the usual quality of your erections during the past 4 weeks" on the EPIC-26 questionnaire
* Agrees to use a condom and another effective method of birth control if he is having sex with a woman of childbearing potential (defined as a premenopausal female capable of becoming pregnant) OR agrees to use a condom if he is having sex with a woman who is pregnant while on study drug and for 3 months following the last dose of study drug. It is recommended that men who have had a vasectomy more than a year prior to trial registration use a condom. Must also agree not to donate sperm.
* Ability to understand and comply with study procedures for the entire length of the study as determined by the site investigator or protocol designee
* Written informed consent and HIPAA authorization for release of personal health information prior to registration. Note: HIPAA authorization may be included in the informed consent or obtained separately. Subject must have the ability to understand and willingness to sign the written informed consent document.
* Ability to swallow pills.
* For patients in whom SBRT/combination RT stratification is pre-specified, prostate volume as determined by MRI, CT, or ultrasound to be less than 90 cc.

Exclusion Criteria:

* Prior surgical, cryotherapy, or high-intensity focused ultrasound for prostate cancer
* Prior orchiectomy or hormonal therapy (gonadotropin releasing hormone (GnRH) agonists, non-steroidal anti-androgens)
* Prior treatment with a first generation AR inhibitor (e.g. bicalutamide, flutamide, nilutamide, cyproterone acetate) or second generation AR inhibitor (e.g.Enzalutamide, Apalutamide, or Darolutamide)
* Prior treatment with other investigational AR inhibitors, CYP17 enzyme inhibitor such as abiraterone acetate, TAK-700, or oral ketoconazole longer than 28 days
* Prior use of estrogens; patients who have used testosterone injections must have ceased utilization within 90 days prior to screening testosterone. Patients who have used any other type of testosterone supplementation (e.g. patches) must have ceased utilization within 45 days prior to screening testosterone.
* Use of 5-α reductase inhibitors (finasteride, dutasteride) within 28 days of randomization.
* Prior radiation therapy that would result in overlap of current radiation therapy fields
* Prior chemotherapy for prostate cancer
* Clinically positive lymph nodes by imaging, sampling, or dissection. Patients with lymph nodes greater than 1.5 cm on short axis will require a negative biopsy for eligibility.
* Metastatic disease, as assessed by abdominal or pelvic computed tomography (CT) or other imaging modality. Patients with 3 intermediate risk factors will require a CT abdomen/pelvis and a bone scan or PET imaging (PSMA PET/CT, fluciclovine PET/CT, etc.).
* Erectile aids other than oral phosphodiesterase (PDE)-5 inhibitors
* History of any of the following: Severe or unstable angina, myocardial infarction, symptomatic congestive heart failure New York Heart Association (NYHA) class III or IV, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), clinically significant ventricular arrhythmias, moderate or severe hepatic impairment (Child Pugh Class B or C), viral hepatitis, or human immunodeficiency virus within 6 months prior to randomization.
* Current untreated hypertension (systolic >= 160 mmHg or diastolic >= 100 mmHg). Patients with one blood pressure reading with systolic < 160 mmHg and diastolic < 100 mmHg within 90 days of registration would be eligible for study.
* Individuals with a history of another malignancy are not eligible if:

  * The cancer is under active treatment
  * The cancer can be seen on radiology scans
  * If they are off cancer treatment, but in the opinion of their oncologist, have a high risk of relapse within 5 years.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drugs
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (NCI-CTCAE version 5.0 Grade 2), psychiatric illness or social situations that would limit compliance with study requirement
* Any condition that, in the opinion of the site investigator, would preclude participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with a PSA nadir <= 0.5 | 6 months from end of treatment
  A response is defined as a PSA nadir <= 0.5 within 6 months from end of treatment

SECONDARY OUTCOMES:
The percentage of patients with good erectile function at 3 months from end of treatment | 3 months from end of treatment
  Good erectile function is defined as firm enough for masturbation or foreplay' or 'firm enough for intercourse' responses to the question "How would you describe the usual quality of your erections during the past 4 weeks" on the EPIC-26 questionnaire.
PSA progression free survival | 3 years
  PSA progression-free survival is defined as the time from randomization to PSA progression (PSA rise of 2 ng/mL above the nadir value).
Metastasis free survival | 3 years
  Metastasis-free survival is defined as the time from randomization to distant metastasis (including bony or visceral) identified on imaging or pathologically, or death due to any cause, or censored at date last known alive.
Cause specific survival | 3 years
  Cause specific survival is defined as the interval from the date of randomization to the date of last known follow-up alive, or the date of death from each of the following causes: prostate cancer, cardiovascular disease, other causes
To evaluate differences in long-term maintenance of erectile function | 3 years
  The answers to EPIC-26 question "How would you describe the usual quality of your erections during the past 4 weeks" from treatment start to the end of follow up at three years show how erectile function has been affected over time.
Rate of Toxicity | 3 years
  Toxicity as measured by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Quality of Life impact as measured by Expanded Prostate Cancer Index (EPIC)-26 | 3 years
  EPIC-26 is a shortened version of the EPIC questionnaire that evaluates subject's urinary incontinence, urinary irritation/obstruction, bowel, sexual, and hormonal domains. EPIC is a robust prostate-cancer health-related QOL instrument that measures a broad spectrum of symptoms and has been widely validated. For each domain, scales range between 0 (worse) and 100 (better).
Global health impact as measured by Patient-Reported Outcome Measurement Information System (PROMIS) Global Health Score | 3 years
  PROMIS is a standardized method for measuring an individual's global health in terms of physical and mental functioning. Scores range from 23.4 (worse) to 63.3 (better).
Memory as measured by the St. Louis University Mental Status Examination (SLUMS) | 3 years
  SLUMS is a single-page exam that measures mild cognitive changes. Scores can be divided as 0-20 (mild dementia), 21-26 (mild cognitive disorder), and 27-30 (normal).
Quality of Life impact as measured by Patient-Reported Outcome Measurement Information System (PROMIS) Sexual Function and Satisfaction Measures (SexFS) Brief Profile Version 2.0. | 3 years
  The PROMIS SexFS Brief Profile v2.0 measures a range of sexual activities, symptoms, functioning, and evaluation of experiences over the past 30 days. Scores range from 31.6 (worse) to 62.7 (better).
Testosterone kinetics | 3 years
  For arm 1, time to Testosterone Recovery is defined as the time from randomization to the date at which the testosterone level returns to a normal level on the assay used, or censored at date of last disease evaluation for those whose testosterone has not reached a normal level. Furthermore, testosterone levels will be compared between arms 1 and 2 at EOT and yearly intervals after EOT.
Cardiovascular events | 3 years
  Time to cardiovascular event is defined as the time from randomization to the date at which the first cardiovascular event occurs. Censoring occurs at date of last disease evaluation for those who did not have a cardiovascular event. Cardiovascular events consisting of myocardial infarction, stroke, deep venous thrombosis, or pulmonary embolism will be collected during study visits and follow-ups.
Time to re-initiation of ADT | 3 years
  Time to re-initiation of ADT is defined as the time from randomization to the date at which ADT is reinitiated. Censoring occurs at date of last disease evaluation for those who are not restarted on ADT.

CONTACTS AND LOCATIONS:
Overall Officials: Martin T. King, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (11):
- United States (11):
  - Stamford Hospital, Stamford, Connecticut
  - Beth Israel Deaconness Medical Center, Boston, Massachusetts
  - Brigham and Women Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center at Milford Regional Medical Center, Milford, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center in Clinical Affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - XCancer Omaha / Urology Cancer Center, Omaha, Nebraska
  - NYU Long Island, Garden City, New York
  - NYU Langone Health, New York, New York
  - Associated Medical Professionals of NY, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Boston Children's Hospital (BCH) - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email tido@childrens.harvard.edu Beth Israel Deaconess Medical Center (BIDMC) - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu Brigham and Women's Hospital (BWH) - Contact the Partners Innovations team at http://www.partners.org/innovation Dana-Farber Cancer Institute (DFCI) - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu Massachusetts General Hospital (MGH) - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Roy A, Green O, Brenneman R, Bosch W, Gay HA, Michalski JM, Baumann BC. Assessing Inter-Fraction Changes in The Size and Position of The Penile Bulb During Daily MR-Guided Radiation Therapy to The Prostate Bed: Do We Need to Adjust How We Plan Radiation in The Post-Radical Prostatectomy Setting to Reduce Risk of Erectile Dysfunction? Clin Genitourin Cancer. 2022 Jun;20(3):e227-e232. doi: 10.1016/j.clgc.2022.01.006. Epub 2022 Jan 11. PMID 35153154